CLINICAL TRIAL: NCT05060874
Title: Comparison of Gripstrength Assessment Between the Gripwise® and JAMAR® Dynamometers in Elderly Inpatients
Brief Title: Gripwise® Versus JAMAR®
Acronym: HANDGAGES
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Bérengère, MD, University Hospital, Caen
Other Study IDs: 2021-A00927-34
Record Dates: First submitted 2021-09-22; First posted 2021-09-29 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Age-Related Sarcopenia
Keywords: aged; inpatients; hand strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single group: gripwise or jamar will be randomly assessed first

SUMMARY:
It is recommended to screen ageing patients for sarcopenia, due to the increased risk of morbimortality if detected positive. According to the consensus of the European Working Group on Sarcopenia in Older People, the diagnosis of sarcopenia is based, among other things, on grip strength measurement.

Our study will compare the performance of the new GRIPWISE digital device with the mechanical dynamometer JAMAR, the gold standard currently used to assess the grip strength. We propose to evaluate it in an elderly hospitalized population where the prevalence of sarcopenia is likely to be high due to the high prevalence of various chronic illness, notably oncological and cardiological ones.

This cross-sectional study will include 348 patients.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 65 or over
* affiliated to a health insurance
* Francophone.

Exclusion Criteria:

* - refusal to participate
* unable to communicate
* unable to use both hands (dominant and non-dominant)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: aged inpatients hospitalized in CAEN University Hospital
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Comparison between Jamar® and Gripwise® values for grip strength measurement | day1
  Intra-class correlation between the best values obtained with each device

SECONDARY OUTCOMES:
comparison according to the patient's position | day1
  correlations of dynamometer measurements between patients assessed in the sitting or lying position
number of attempt to reach the maximum value | day1
  Comparison of the three measurements obtained for each patient with each device
factors influencing detected weakness | day1
  significant difference in the rate of women detected as weak with a handgrip <16kg and men <27kg, between the different reasons for hospitalisation, the number of days of hospitalisation, and between the different chronic cancerous and non-cancerous pathologies (Updated Charlson Comorbidity Index), the age groups 65-79 years and ≥80 years
satisfaction using the devices | day1
  rate of patients finding one of both device easier to use

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère Beauplet, MD, Principal Investigator — Caen UH
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided